CLINICAL TRIAL: NCT01097382
Title: National, Multicenter, Open Label, Phase IV, Before-after Design Study, in Adult Patients With Primary Insomnia to Evaluate Sleep Satisfaction and Psychomotor Performance After 1 Month of Treatment With Zolpidem CR (Ambien®CR) in 6 Sites in Argentina
Brief Title: Sleep Satisfaction and Psychomotor Performance of Adults
Acronym: MORFEO CR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZOLPI_L_04551; U1111-1116-9105 (Other: UTN)
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Sleep Disorders
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Zolpidem

ARMS (1):
- AMBIEN CR (Experimental): AMBIEN CR 12.5 mg once daily immediately before bedtime or in elderly/hepatically impaired patients: 6.25 mg once daily immediately before bedtime
  Interventions: Drug: ZOLPIDEM

INTERVENTIONS:
Drug: ZOLPIDEM — Pharmaceutical form: tablet Route of administration: oral Dose regimen: once daily

SUMMARY:
Primary Objective:

To assess sleep satisfaction before and after Zolpidem CR (Ambien CR) administration

Secondary Objective:

To assess Psychomotor Performance before and after Zolpidem CR (Ambien CR) administration

ELIGIBILITY:
Inclusion criteria:

* Patients consulting Psychiatrists (private or hospital) -whatever the reason for consulting- who present with chronic primary insomnia from the DSM IV (Diagnostic and Statistical Manual - Revision 4).
* Accepting to participate in the study and signing informed consent

Exclusion criteria:

* Pregnancy or breastfeeding.
* Current severe neuropsychiatric disorder (i.e. psychosis, obsessive compulsive disorder, major depression, dementia of Alzheimer or vascular type) according to DSM IV criteria.
* History of substance abuse or dependence (including alcohol) within the past year.
* Hypersensitivity to zolpidem or its excipients.
* Severe hepatic insufficiency
* Severe and/or acute respiratory insufficiency
* Myasthenia gravis.
* OTC (Over The Counter) sleep remedies or prescription sleep medications within 2 weeks or 5 half-life before screening.
* Severe medical illness.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Sleep satisfaction score (LSEQ = Leeds sleep evaluation questionnaire) | at Baseline, at V2 (26 +/- 2 days)

SECONDARY OUTCOMES:
Psychomotor Performance (DSST / Digit Symbol Substitution Test and ESS / Epworth Sleepiness Scale) | at Baseline, at V2 (26 +/- 2 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- Argentina (6):
  - Investigational Site Number 10, Buenos Aires
  - Investigational Site Number 1, C.a.b.a.
  - Investigational Site Number 4, C.a.b.a.
  - Investigational Site Number 6, C.a.b.a.
  - Investigational Site Number 2, Capital Federal
  - Investigational Site Number 3, La Plata